CLINICAL TRIAL: NCT04912193
Title: Low Preoperative Antithrombin III Level is Associated With Postoperative Acute Kidney Injury After Liver Transplantation
Brief Title: Antithrombin III and Post-liver Transplantation Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kyoung-Sun Kim, Senior Clinical Fellow, Asan Medical Center
Other Study IDs: 2019-1699
Record Dates: First submitted 2021-05-30; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Liver Transplantation and Antithrombin
Keywords: acute kidney injury; antithrombins; liver transplantation
MeSH Terms: conditions — Acute Kidney Injury | interventions — Antithrombin III

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- antithrombin III < 50 %: preoperative antithrombin III levels <50%
  Interventions: Drug: Antithrombin III
- Antithrombin III ≥ 50 %: preoperative antithrombin III levels ≥ 50 %

INTERVENTIONS:
Drug: Antithrombin III — In liver transplant recipients with baseline antithrombin III levels lower than 50%, exogenous Antithrombin III was administrated during the anhepatic phase of the liver transplant surgery.
  Groups: antithrombin III < 50 %

SUMMARY:
The reno-protective effect of Antithrombin III (ATIII) has been well-studied in various animal studies; however, little is known about the effect of ATIII on kidney function in patients undergoing liver transplantation (LT). This study aimed to determine the association between preoperative ATIII level and postoperative acute kidney injury (AKI) after LT (post-LT AKI).

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent either living- or deceased-donor LT (LDLT, DDLT) from January 2010 to January 2018

Exclusion Criteria:

* patients who underwent re-transplantation
* patients who were previously diagnosed with end-stage renal disease or Chronic kidney disease
* patients who were being treated with continuous renal replacement therapy
* preoperative or postoperative Antithrombin III levels were not available

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who underwent either living- or deceased-donor LT (LDLT, DDLT) from January 2010 to January 2018 in Asan Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 2395 (Actual)
Dates: Start 2010-01-04 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | postoperative 7 day
  serum creatinine >0.3 mg/dL within POD 2 or increase by >1.5 times within POD 7 according to the criteria set by the Kidney Disease: Improving Global Outcomes (KDIGO) classification

SECONDARY OUTCOMES:
chronic kidney disease | postoperative 3 months
  glomerular filtration rate less than 60 mL∙min-1∙1.73m-2 on two consecutive occasions at least 3 months apart
early allograft dysfucion | postoperative 7 day
  at least one of the following: total bilirubin ≥10 mg/dL on postoperative day (POD) 7, prothrombin time (INR) ≥1.6 on POD 7, and alanine or aspartate aminotransferases >2000 IU/L within POD 7

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Levy JH, Sniecinski RM, Welsby IJ, Levi M. Antithrombin: anti-inflammatory properties and clinical applications. Thromb Haemost. 2016 Apr;115(4):712-28. doi: 10.1160/TH15-08-0687. Epub 2015 Dec 17. PMID 26676884
- [Background] Wu R, Kong Y, Yin J, Liang R, Lu Z, Wang N, Zhao Q, Zhou Y, Yan C, Wang F, Liang M. Antithrombin Ⅲ is a Novel Predictor for Contrast Induced Nephropathy After Coronary Angiography. Kidney Blood Press Res. 2018;43(1):170-180. doi: 10.1159/000487499. Epub 2018 Feb 16. PMID 29466798
- [Background] Lu Z, Cheng D, Yin J, Wu R, Zhang G, Zhao Q, Wang N, Wang F, Liang M. Antithrombin III Protects Against Contrast-Induced Nephropathy. EBioMedicine. 2017 Mar;17:101-107. doi: 10.1016/j.ebiom.2017.02.009. Epub 2017 Feb 12. PMID 28219627
- [Result] Wang F, Zhang G, Lu Z, Geurts AM, Usa K, Jacob HJ, Cowley AW, Wang N, Liang M. Antithrombin III/SerpinC1 insufficiency exacerbates renal ischemia/reperfusion injury. Kidney Int. 2015 Oct;88(4):796-803. doi: 10.1038/ki.2015.176. Epub 2015 Jun 24. PMID 26108065
- [Result] Yin J, Wang F, Kong Y, Wu R, Zhang G, Wang N, Wang L, Lu Z, Liang M. Antithrombin III prevents progression of chronic kidney disease following experimental ischaemic-reperfusion injury. J Cell Mol Med. 2017 Dec;21(12):3506-3514. doi: 10.1111/jcmm.13261. Epub 2017 Aug 2. PMID 28767184